CLINICAL TRIAL: NCT02433691
Title: Simultaneous Aerobic Exercise and Memory Training in Older Adults With Subjective Memory Complaints
Brief Title: Memory and Exercise Training Study in Older Adults With Subjective Memory Complaints
Acronym: MET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Merrill, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, David Merrill, MD, PhD, Assistant Clinical Professor, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 14-001411
Record Dates: First submitted 2015-04-13; First posted 2015-05-05 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Memory Impairment
Keywords: (An)aerobic exercise; memory training; cognitive benefits
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sequential Exercise and Memory Training (Active Comparator): Aerobic exercise via stationary bicycling followed by memory training.
  Interventions: Other: sequential aerobic exercise
- Simultaneous Exercise & Memory Training (Experimental): Simultaneous aerobic exercise via stationary bicycling while receiving memory training.
  Interventions: Other: simultaneous aerobic exercise
- Stretching and Toning (Placebo Comparator): Anerobic stretching and toning followed by memory training
  Interventions: Other: stretching and toning

INTERVENTIONS:
Other: simultaneous aerobic exercise — stationary bicycling at 65% of heart rate reserve for 30 minutes while receiving memory training.
  Arms: Simultaneous Exercise & Memory Training
Other: sequential aerobic exercise — stationary bicycling at 65% of heart rate reserve for 30 minutes followed by memory training.
  Arms: Sequential Exercise and Memory Training
Other: stretching and toning — anaerobic stretching and toning followed by memory training.
  Arms: Stretching and Toning

SUMMARY:
This pilot study is a first step in a rapidly growing area of clinical research to create the most effective means to combat age-related losses in cognitive function through preventive lifestyle strategies such as physical exercise and memory training. This study will develop innovative simultaneous exercise and memory training programs in non-demented volunteers with subjective memory complaints (controls or MCI). Our primary goal is to assess the cognitive impact of 4-week memory training programs done twice weekly: 1. during simultaneous aerobic exercise (SIM-AR-MET), 2. sequentially after aerobic exercise (SEQ-AR-MET), or 3. without aerobic exercise (replaced with sequential stretching and toning) (SEQ-ST-MET). The investigators will also measure potential metabolic (e.g., glucose, lipid panel) and molecular (serum BDNF) mediators of observed cognitive changes in a subset of participants (those at the UCLA CTRC/IPCN site).

DETAILED DESCRIPTION:
A total of 90 non-demented healthy older adult volunteers (age 60-75) with subjective memory complaints (controls or MCI) will be screened and enrolled into the study. The CTRC/IPCN site will enroll 30 subjects (10 in each group); the MPTF site will enroll 60 subjects (20 in each group). Baseline assessments will include neuropsychological testing of all study subjects. At UCLA CTRC/IPCN, baseline assessments will also include cardiorespiratory fitness, body composition, YMCA fitness tests, and blood-based markers of metabolism and plasticity. To control for total activity levels, all study subjects will wear continuous physical activity monitors (FitBit accelerometers) and keep exercise and cognitive activity logs during the entire study. All subjects (n = 90) will first complete a 1-week observational period to capture baseline activity levels. Subjects will then be randomized to one of three groups: SIM-AR-E&MT, SEQ-AR-E&MT, or SEQ-ST-MET (n = 30 per group). SIM-AR-MET and SEQ-AR-MET subjects will complete a 3-week exercise only 'ramp-up' period consisting of twice weekly 1-hour sessions practicing stationary bicycling, improving cardiovascular fitness enough to complete the upcoming 4-weeks of MET sessions (described below), and practicing stretching and toning; SEQ-ST-MET subjects 3-week exercise only 'ramp-up' period will consist of an equal number of six stretching and toning sessions (no aerobic components). All 3 programs will then have two 2-hour sessions per week for 4 weeks. The SIM-AR-MET and SEQ-ST-MET subjects will do stretching/toning during the first hour; SEQ-AR-MET subjects will do aerobic cycling during the first hour. During the second half of the sessions, all 3 groups will first learn new memory training strategies while sedentary. SIM-AR-MET subjects will then practice the memory techniques while cycling while SEQ-AR-MET and SEQ-ST-MET subjects will practice the memory techniques while still sedentary. The three groups will have group specific exercise and memory training homework assignments, along with monitoring of activity and logging of cognitively enriching activities. The NP testing will be done again at the end of the 4 weeks of memory training classes for all study subjects. UCLA CTRC/IPCN subjects will have the additional testing done at baseline (e.g., blood-based markers, etc.).

Consideration was given to having a purely observational 'wait-list' group, but in our experience with this population such groups have typically initiated greater levels of self-guided exercise and memory training in reaction to being put on a wait list. Alternatively, if no increase in activity or memory training is undertaken by wait list subjects, the investigators would not expect any differences in cognitive performance to be measurable within the brief 3 month total time frame of this initial study. The investigators also considered have a group do aerobic exercise immediately after memory training, but based on current literature, this combination seemed the least likely to impact memory synergistically. Thus, these two groups will be deferred for the pilot until later, larger studies can be done to confirm or refute these hypotheses. Similarly, while our primary aim assessing change in NP performance will be tested in all subjects, the pilot nature of the study prohibits testing of secondary aims in both sites. The academic medical center site will leverage the assistance of the UCLA CTRC/IPCN to accomplish preliminary testing of the secondary aims in 30 subjects, while the UCLA MPTF community site will test only the primary study aim of change in NP performance.

ELIGIBILITY:
Inclusion Criteria:

* In good health
* Have memory problems or complaints
* Living independently

Exclusion Criteria:

* History of neurodegenerative disease or dementia
* Major psychiatric conditions
* Neurological disorders
* Active alcohol or substance abuse
* Head trauma or systemic diseases affecting brain function
* Uncontrolled hypertension or cardiovascular disease

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Effects of the MET interventions on cognition (comparing baseline vs. end-of-study NP testing) | up to 9 months
  Change from baseline in composite measure of memory related tasks including retention, attention, and mood.

SECONDARY OUTCOMES:
Changes in BDNF levels in response to the interventions | up to 9 months
  Increase of baseline measurement for BDNF levels.
Physical health measures | up to 9 months
  Change in baseline in composite measurement of weight (loss), and increase in physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah McEwen, Ph.D., Principal Investigator — UCSD
Locations (1):
- UCLA Longevity Center, Los Angeles, California, United States

REFERENCES:
- [Result] Miller KJ, Siddarth P, Gaines JM, Parrish JM, Ercoli LM, Marx K, Ronch J, Pilgram B, Burke K, Barczak N, Babcock B, Small GW. The memory fitness program: cognitive effects of a healthy aging intervention. Am J Geriatr Psychiatry. 2012 Jun;20(6):514-23. doi: 10.1097/JGP.0b013e318227f821. PMID 21765343
- [Result] Barnes DE, Yaffe K, Satariano WA, Tager IB. A longitudinal study of cardiorespiratory fitness and cognitive function in healthy older adults. J Am Geriatr Soc. 2003 Apr;51(4):459-65. doi: 10.1046/j.1532-5415.2003.51153.x. PMID 12657064
- [Result] Erickson KI, Miller DL, Roecklein KA. The aging hippocampus: interactions between exercise, depression, and BDNF. Neuroscientist. 2012 Feb;18(1):82-97. doi: 10.1177/1073858410397054. Epub 2011 Apr 29. PMID 21531985
- [Result] Goodwin VA, Richards SH, Taylor RS, Taylor AH, Campbell JL. The effectiveness of exercise interventions for people with Parkinson's disease: a systematic review and meta-analysis. Mov Disord. 2008 Apr 15;23(5):631-40. doi: 10.1002/mds.21922. PMID 18181210
- [Result] Hillman CH, Erickson KI, Kramer AF. Be smart, exercise your heart: exercise effects on brain and cognition. Nat Rev Neurosci. 2008 Jan;9(1):58-65. doi: 10.1038/nrn2298. PMID 18094706
- [Result] Petzinger GM, Fisher BE, McEwen S, Beeler JA, Walsh JP, Jakowec MW. Exercise-enhanced neuroplasticity targeting motor and cognitive circuitry in Parkinson's disease. Lancet Neurol. 2013 Jul;12(7):716-26. doi: 10.1016/S1474-4422(13)70123-6. PMID 23769598
- [Result] Barnes DE, Santos-Modesitt W, Poelke G, Kramer AF, Castro C, Middleton LE, Yaffe K. The Mental Activity and eXercise (MAX) trial: a randomized controlled trial to enhance cognitive function in older adults. JAMA Intern Med. 2013 May 13;173(9):797-804. doi: 10.1001/jamainternmed.2013.189. PMID 23545598
- [Result] Oswald WD, Rupprecht R, Gunzelmann T, Tritt K. The SIMA-project: effects of 1 year cognitive and psychomotor training on cognitive abilities of the elderly. Behav Brain Res. 1996 Jun;78(1):67-72. doi: 10.1016/0166-4328(95)00219-7. PMID 8793039
- [Result] Berchtold NC, Castello N, Cotman CW. Exercise and time-dependent benefits to learning and memory. Neuroscience. 2010 May 19;167(3):588-97. doi: 10.1016/j.neuroscience.2010.02.050. Epub 2010 Feb 26. PMID 20219647
- [Result] Rasmussen P, Brassard P, Adser H, Pedersen MV, Leick L, Hart E, Secher NH, Pedersen BK, Pilegaard H. Evidence for a release of brain-derived neurotrophic factor from the brain during exercise. Exp Physiol. 2009 Oct;94(10):1062-9. doi: 10.1113/expphysiol.2009.048512. Epub 2009 Aug 7. PMID 19666694
- [Derived] McEwen SC, Siddarth P, Rahi B, Kim Y, Mui W, Wu P, Emerson ND, Lee J, Greenberg S, Shelton T, Kaiser S, Small GW, Merrill DA. Simultaneous Aerobic Exercise and Memory Training Program in Older Adults with Subjective Memory Impairments. J Alzheimers Dis. 2018;62(2):795-806. doi: 10.3233/JAD-170846. PMID 29480182